CLINICAL TRIAL: NCT06377098
Title: Sildenafil Citrate to Improve Maternal and Neonatal Outcomes in Low-Resource Settings: A Randomized Pilot Feasibility Trial: Pilot Randomized Intrapartum Sildenafil in Mothers
Brief Title: Intrapartum Sildenafil in Laboring Mothers
Acronym: PRISM
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Funding not obtained
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University Teaching Hospital, Lusaka, Zambia (Other); Egerton University (Other); Cameroon Baptist Convention Health (Other)
Responsible Party: Principal Investigator, Waldemar A. Carlo, Edwin M. Dixon Professor of Pediatrics, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UAB-300010901; UAB Dixon Endowed Ch/3102800 (Other Grant/Funding Number: UAB Dixon Endowed Chair)
Record Dates: First submitted 2024-04-12; First posted 2024-04-22 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Neonatal Asphyxia; Intrapartum Fetal Distress; Development, Infant; Intrapartum Asphyxia
Keywords: Sildenafil citrate
MeSH Terms: conditions — Asphyxia Neonatorum | interventions — Sildenafil Citrate; Tablets

STUDY DESIGN:
Intervention Model Description: Double blinded, placebo-controlled, 1:1 parallel allocation, randomized feasibility trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The only person who will be unmasked will be the pharmacist who will dispense the study medication--either sildenafil 50mg or identical placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Sildenafil 50mg (Active Comparator): Sildenafil citrate 50mg given orally every eight hours up to 3 doses while mother is in labor
  Interventions: Drug: Sildenafil 50 mg Oral Tablet
- Placebo (Placebo Comparator): Identical-appearing treatment that does not contain the test drug given orally every eight hours up to 3 doses while mother is in labor
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Sildenafil 50 mg Oral Tablet — Sildenafil 50 mg given orally every eight hours up to three times while mother is in labor
  Other Names: Revatio; Sildenafil
  Arms: Oral Sildenafil 50mg
Drug: Placebo Oral Tablet — Placebo table given orally every eight hours up to three times while mother is in labor
  Arms: Placebo

SUMMARY:
The goal of this feasibility pilot clinical trial is to learn if sildenafil citrate 50mg orally, up to three times during labor, can be appropriately administered, with limited clinical side effects, to laboring mothers to determine feasibility across a spectrum of available healthcare resources.

The main questions it aims to answer are:

* What are the fetal heart rate monitoring practices in a low-resource setting?
* What are the indications for operative delivery in a low-resource?
* What is the rate of relevant primary and secondary outcomes to possibly target in a large RCT of intrapartum sildenafil?
* What is the limited effect size of sildenafil citrate on maternal and neonatal outcomes in a low-resource setting?

Researchers will compare the administration of sildenafil citrate 50 mg orally to a placebo (a look-alike substance that contains no drug) to see if procedures are feasible, the drug is tolerated, the target outcomes are achievable, and effect size is as expected.

Participants will:

* Take Sildenafil 50 mg/placebo every eight hours or a placebo every eight hours for up to 24 hours during labor
* Have the (mothers & babies) medical charts reviewed for outcomes, including fetal distress, operative delivery, maternal side effects, neonatal bag & mask ventilation, Apgar scores, and seizures.
* Have a neonatal neurological assessment prior to discharge
* Have phone call assessments for re-hospitalization or mortality 7 days post-delivery
* Receive child development assessments at 1 year, 2 years and 3 years of age by the Ages and Stages Questionnaire administered via a telephone call

The results of this feasibility pilot trial will be used to inform the design and conduct of a large pragmatic randomized controlled trial to determine if sildenafil citrate, compared to placebo, will decrease fetal distress and perinatal asphyxia.

DETAILED DESCRIPTION:
After informed consent obtained, mother will be randomized, using computer-generated stratified randomization codes by the pharmacy. Clinicians, researcher, and primary caregivers will be masked. Subjects will be randomly assigned to either the treatment arm or the placebo concurrent control.

Eligible women who consent for the study will be randomized to receive sildenafil 50 mg orally every 8 hours up to a total of 3 doses or to receive the placebo every 8 hours up to a total of 3 does during the course of labor. Neither medication no placebo will be given following completion of labor. All additional care of the mother and infant will be provided according to the local standard of care. Outcomes will be collected following delivery, discharge, and 7-days post-partum. 7-day follow-up for outcomes will be obtained per a telephone call. One, two, and three year infant developmental and behavior outcome will be assessed using the Ages and Stages Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women presenting in early labor with a term pregnancy (≥ 37 weeks gestation)

   * Early labor will be defined as cervical dilation less than or equal to 6 cm
   * Gestational age will be calculated from the most reliable variable using the following hierarchy of reliability: 2) gestational dating ultrasound completed at any time during the pregnancy (with preference to the earliest exam); 2) date of last menstrual period if menses are regular.
2. Planned vaginal delivery and admission to health facility with clear plan for spontaneous or induced vaginal delivery
3. Maternal age ≥ 18yrs or minors 14-17yrs eligible in countries where married or pregnant minors or their authorized representatives are legally permitted to give consent
4. A single, live fetus in cephalic presentation confirmed prior to randomization

Exclusion Criteria:

1. Unknown gestational age
2. Maternal history of cesarean delivery
3. Advanced stage of labor (>6 cm or 10 cm cervical dilation per local standards) and pushing, or too distressed to understand, confirm, or give informed consent regardless of cervical dilation
4. Not capable of giving consent due to other health problems, such as obstetric emergencies (i.e. antepartum hemorrhage) or mental disorder
5. Maternal contraindication to sildenafil therapy, such as hypersensitivity to nitrates or nitrites
6. Any medical condition considered a contraindication per the judgement of site investigators
7. Recognized fetal anomaly
8. Any maternal medical condition or status that precludes informed consent
9. Non-emancipated minors (as per local regulations
10. Plan for cesarean delivery prior to enrollment
11. Previous randomization in the trial

Ages: 0 Days to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of perinatal mortality | 96 hours after enrollment
  Documentation of stillbirth or neonatal death
Percentage of operative delivery | 96 hours after enrollment
  Documentation of type of delivery
Indication for operative delivery | 96 hours after enrollment
  Documentation of type of delivery

SECONDARY OUTCOMES:
Percentage of mothers who received fetal heart rate monitoring | 96 hours after enrollment
  Documentation of rate of heart rate monitoring
Indication for fetal heart rate monitoring | 96 hours after enrollment
  Documentation of the indication for use of fetal heart rate monitoring
Apgar Score | 1 minute and 5 minutes after birth
  Documentation of Apgar score at 1 minute and 5 minutes (Value 0-10, with 10 meaning better outcome)
Percentage of use of bag and mask ventilation in neonates | 20 minutes after delivery
  Documentation of the use of bag and mask ventilation as resuscitation after delivery
Percentage of neonates with neonatal encephalopathy | 24 hours after birth
  Documentation of neonatal neurological exam determined by "modified Sarnat Score (no, mild, moderate, and severe)" ; higher score indicates more severe encephalopathy
Percentage of neonates with neonatal encephalopathy | 24 hours after birth
  Documentation of neonatal neurological exam determined by "Thompson Score (no, mild, moderate and severe)"; higher score indicates more severe encephalopathy
Percentage of neonates with hypoxemia | 48 hours after birth or at discharge, if early discharge
  Documentation of saturations < 95% measured by noninvasive pre/post pulse oximetry
Percentage of infants with neonatal hypoxic-ischemic encephalopathy | 96 hours after enrollment
  Documentation of neonatal encephalopathy
Percentage of neonatal ICU admissions | 96 hours after enrollment
  Documentation of admission to the Neonatal Intensive Care Unit or comparable level of care
Percentage of maternal rehospitalization | 7 days
  Maternal rehospitalization after initial discharge from the hospital assessed by telephone call to mother
Percentage of neonatal rehospitalization | 7 days
  Neonatal rehospitalization after initial discharge from the hospital assessed by telephone call to mother
Infant/child developmental assessment | 12 months, 24 months, 36 months
  Score on "Ages and Stages Questionnaire" obtained by telephone call to parent (developmental assessment tool which scores items (Yes=10, Sometimes=5, Not Yet=0) in areas of Communication, Gross Motor, Fine Motor, Problem Solving, and Personal-Social. Scoring of items are totaled and placed on a graph indicating cutoff score. If score is above cutoff, the child's development appears to be on schedule; near the cutoff, may provide learning activities and monitor; and below cutoff, requiring further assessment. 12-month cutoffs (Communication 15.64; Gross Motor 21.49; Fine Motor 34.50; Problem Solving 27.32 and Personal-Social 21.73); 24-month cutoffs ((Communication 25.17; Gross Motor 38.07; Fine Motor 35.16; Problem Solving 29.78 and Personal-Social 31.54); and 36-month cutoffs (Communication 30.99; Gross Motor 36.99; Fine Motor 18.07; Problem Solving 30.29 and Personal-Social 35.33)

CONTACTS AND LOCATIONS:
Overall Officials: Waldemar A Carlo, MD, Principal Investigator — University of Alabama at Birmingham
Locations (3):
- Cameroon Baptist Convention Health Services, Douala, Cameroon
- Egerton University/Nakuru County Referral Hospital, Nakuru, Kenya
- University Teaching Hospital, Lusaka, Zambia